CLINICAL TRIAL: NCT02128126
Title: A Multicenter, Open Label Phase I/II Study to Determine the Safety and Immune Modulating Effects of the Therapeutic Human Papilloma Virus 16 (HPV16) E6/E7 Long Peptides Vaccine (ISA101/ISA101b) Immunotherapy in Combination With Standard of Care Therapy (Carboplatin and Paclitaxel With or Without Bevacizumab) in Women With HPV16 Positive Advanced or Recurrent Cervical Cancer Who Have no Curative Treatment Options
Brief Title: Study of the Therapeutic Vaccine (ISA101/ISA101b) to Treat Advanced or Recurrent Cervical Cancer
Acronym: CervISA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ISA Pharmaceuticals (Industry)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISA-HPV-01-12; 2013-001804-12 (EudraCT Number)
Record Dates: First submitted 2014-04-18; First posted 2014-05-01 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Cervical Cancer
Keywords: Advanced or recurrent cervical cancer; HPV16 positive; No curative treatment options
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ISA101/ISA101b (Experimental): The maximum total treatment duration for a patient is six cycles (1 cycle is 21 days) for a total of 18 weeks. On day 15 of cycles 2, 3 and 4 patients are to receive the vaccination scheme of ISA101/ISA101b. Patients will be vaccinated with a fixed dose of ISA101/ISA101b every three weeks for a total of three rounds of vaccination. Four dose levels of ISA101 have been tested. ISA101b will be tested in bridging cohorts.
  Interventions: Drug: ISA101/ISA101b

INTERVENTIONS:
Drug: ISA101/ISA101b — Four dose levels ISA101/ISA101b
  Other Names: HPV Type 16 E6/E7 Synthetic Long Peptides Vaccine

SUMMARY:
The purpose of the study is to assess the safety, tolerability and the HPV-specific immune responses of different doses of ISA101 vaccine with or without pegylated IFNα as combination therapy with carboplatin and paclitaxel.

To qualitatively assess the safety profile and the HPV-specific immune responses of ISA101b vaccine compared to ISA101 at the same dose levels.

To assess the safety and the HPV-specific immune responses of ISA101b vaccine with carboplatin, paclitaxel with or without bevacizumab.

DETAILED DESCRIPTION:
A majority of cervical carcinomas are caused by an uncontrolled, persistent infection with high risk Human Papilloma Virus (HPV). ISA101/ISA101b is a novel therapeutic synthetic long peptide (SLP) vaccine targeting HPV16 which is being developed and has shown efficacy in patients with high-grade premalignant vulvar lesions caused by HPV with only minor toxicity. For most advanced cancers, chemotherapy remains the treatment modality of choice but has been considered to be immunosuppressive. However, accumulating evidence indicates that many modalities of conventional chemotherapy not only are less immunosuppressive than previously thought but in fact can exert favorable effects on the tumor micro-environment by interfering with suppressive immune cells and by stimulating the release of immune activating molecules by tumor cells. Thus chemotherapy may enhance tumor-specific immunity and synergize with cancer immunotherapy. Addition of pegylated interferon alpha (IFNα) two-b (IIb) to vaccination might even further improve the immune response. This multicenter, open label, non-randomized Phase I/II study will be performed to assess the safety and tolerability of the ISA101/ISA101b vaccine, and the immune modulating effects of ISA101 (with or without pegylated IFNα)/ISA101b when combined with carboplatin and paclitaxel, with or without bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥ 18 years of age.
2. Cervical cancer confirmed by histology.
3. Advanced or metastatic or recurrent cervical cancer confirmed by clinical and/or radiological proof with no curative treatment options.
4. For cohort 10 (and 12), i.e. patients eligible to receive bevacizumab at each site per standard of care, patients may be primary stage IVB (including persistent) or first recurrent carcinoma of the uterine cervix (squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma). Prior treatment with chemotherapy for recurrent disease is not permitted. However, one prior line of chemotherapy with platinum during primary radio-chemotherapy or platinum-base chemotherapy as neoadjuvant chemotherapy prior to surgery is permitted
5. Tumour must be HPV16 positive.
6. Patients should be eligible for chemotherapy with carboplatin and paclitaxel, and have consented with chemotherapy with carboplatin and paclitaxel, before the start of the informed consent procedure for the study.
7. Performance status (WHO scale/ECOG) 1.
8. Written informed consent according to local guidelines.
9. Written approval by the treating physician/investigator of his/her clinical judgment that the patient has a reasonable life expectancy and is sufficiently fit and motivated to complete the study treatment and comply to all study procedures conform the protocol.

Exclusion Criteria:

Treatment:

1. Prior treatment with anti-HPV agents.
2. Chronic systemic steroid use. Local application (i.e. stable doses of topical or inhaled corticosteroids) is allowed.
3. Less than 4 weeks since the last treatment with other cancer therapies, (i.e. endocrine therapy, immunotherapy, radiotherapy, chemotherapy, etc), less than 8 weeks for cranial radiotherapy, and less than 6 weeks for nitrosoureas and mitomycin C.
4. Toxicities resulting from previous anti-cancer therapy must be resolved to ≤ grade 2.
5. Recent treatment (within 30 days of first study treatment) with another investigational drug.
6. Patients with known hypersensitivity to any component of the Investigational Medicinal Product.
7. Any contraindication to the use of authorized applied products (i.e. paclitaxel, carboplatin or bevacizumab).

   Haematology and biochemistry:
8. Inadequate bone marrow function: Absolute Neutrophil Count (ANC) < 1.5 x 109/L, or platelet count < 100 x 109/L or hemoglobin < 6 mmol/L.
9. Inadequate liver function, defined as:

   * Serum (total) bilirubin > 2 x upper normal limit (ULN);
   * Aspartate Aminotransferase (ASAT) or Alanine Aminotransferase (ALAT) > 2.5 x ULN (> 5 x ULN in patients with liver metastases);
   * Alkaline phosphatase levels > 2.5 x ULN (> 5 x ULN in patients with liver metastases, or > 10 x ULN in patients with bone metastases).

   Other:
10. Clinical suspicion or radiological evidence of brain or leptomeningeal metastases.
11. Previous or current malignancies at other sites, with the exception of basal or squamous cell carcinoma of the skin and with the exception of other malignancies from which the patient may be considered cured as evidenced by complete regression of all lesions >10 years ago.
12. Active HIV, chronic hepatitis B or C infection.
13. Patients of childbearing potential not willing to consistently and correctly us a contraceptive method according to ICH (M3) resulting in low failure rate, i.e. less that 1% per year such as oral contraceptives or use of effective means of contraception.
14. Pregnancy or lactation. Serum pregnancy test to be performed within 7 days prior to study treatment start in patients of childbearing potential.
15. Major surgical procedure within 28 days prior to the first study treatment.
16. Uncontrolled sustained hypertension (systolic > 180 mm Hg and/or diastolic > 110mm Hg).
17. Clinically significant (i.e. active) cardiovascular disease defined as:

    * Stroke within ≤ 6 months prior to day 1;
    * Transient Ischemic Attack (TIA) within ≤ 6 months prior to day 1;
    * Myocardial infarction within ≤ 6 months prior to day 1;
    * Unstable angina;
    * New York Heart Association (NYHA) Grade II or greater Congestive Heart Failure (CHF);
    * Serious cardiac arrhythmia requiring medication;
18. History of severe bronchial asthma and/or severe allergy.
19. Evidence of any other medical conditions that may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-09; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
HPV-specific immune responses | 4 months
  HPV-specific immune responses to different doses of the ISA101 vaccine with or without pegylated interferon alpha (INFα) as combination therapy with carboplatin and paclitaxel will be determined. The HPV-specific immune responses to ISA101b will be qualitatively compared to the responses at the same dose level(s) of ISA101.

SECONDARY OUTCOMES:
Evaluate the clinical efficacy by antitumor efficacy according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | one year

OTHER OUTCOMES:
Evaluate the general responsiveness of the immune system as measured by explorative assays. | 4 months
  General responsiveness of the immune system as measured by explorative assays in particular:
  1. Lymphocyte proliferation
  2. Antigen Presenting Cell (APC) function tests
  3. Assay of myeloid and lymphoid cell composition
  4. Recall proliferative responses of Peripheral Blood Mononuclear Cells(PBMCs) in response to common microbial antigens

CONTACTS AND LOCATIONS:
Overall Officials: Winald Gerritsen, Oncologist, Principal Investigator — Radboud University Medical Center
Locations (15):
- Belgium (5):
  - UZA, Antwerp
  - Chirec Cancer Institute, Brussels
  - UZG, Ghent
  - UZL, Leuven
  - CHU of Liege Site Citadelle, Liège
- Germany (4):
  - Universitätsklinikum Düsseldorf - Frauenklinik, Düsseldorf
  - Universitätsklinikum Essen - Klinik für Frauenheilkunde, Essen
  - Medizinische Hochschule Hannover - Klinik für Frauenheilkunde, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
- Netherlands (6):
  - NKI/AVL, Amsterdam
  - AMC, Amsterdam
  - UMCG, Groningen
  - LUMC, Leiden
  - MUMC, Maastricht
  - Radboud UMC, Nijmegen

REFERENCES:
- [Derived] Domingos-Pereira S, Galliverti G, Hanahan D, Nardelli-Haefliger D. Carboplatin/paclitaxel, E7-vaccination and intravaginal CpG as tri-therapy towards efficient regression of genital HPV16 tumors. J Immunother Cancer. 2019 May 6;7(1):122. doi: 10.1186/s40425-019-0593-1. PMID 31060612